CLINICAL TRIAL: NCT04894396
Title: A Randomised Control Trial Comparing Prefabricated Orthotics With and Without Metatarsal Pad in Decreasing Pain and Fear of Falling in Older Adults
Brief Title: Orthotics, Pain & Fear of Falling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Talita Cumi Ltd. (Industry)
Collaborators: Aetrex Worldwide Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FFPETFETS003
Record Dates: First submitted 2021-05-14; First posted 2021-05-20 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Foot Pain; Foot Functionality; Fear of Falling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prefabricated Orthotics with metatarsal pad (Experimental): Participants in Group A will receive the Orthotic with the metatarsal pad (L 2305) according to participants shoe size (https://www.aetrex.com/search?q=l2305&search-button=&lang=en_US). When the investigators provide the Orthotics, an instruction sheet will also be provided, explaining how to use the orthotic. Alternatively, an online video tutorial on how to use the Orthotic will also be available throughout the study. Participants will be required to use the Orthotic wherever possible for a period of 6 weeks, whilst continuing with usual activities.
  Interventions: Device: Aetrex L2305 Premium Memory Foam Orthotics W/ Metatarsal Support
- Prefabricated Orthotics without metatarsal pad. (Active Comparator): Participants in Group B will receive the neutral Orthotic with a cupped heel (L 2300) according to participants shoe size (https://www.aetrex.com/search?q=l2300&search-button=&lang=en_US). When the investigators provide the Orthotics, an instruction sheet will also be provided, explaining how to use the Orthotic. Alternatively, an online video tutorial on how to use the Orthotic will also be available throughout the study. Participants will be required to use the Orthotic wherever possible for a period of 6 weeks, whilst continuing with usual activities
  Interventions: Device: Aetrex L2300 Premium Memory Foam Orthotics

INTERVENTIONS:
Device: Aetrex L2305 Premium Memory Foam Orthotics W/ Metatarsal Support — An Orthotic insole to be inserted into shoes. Features Aetrex Arch Support to help biomechanically align the body & help prevent common foot pain such as Plantar Fasciitis, Arch Pain and Metatarsalgia. For medium to high arches with forefoot pain, featuring a cupped heel to cushion and stabilize the back of foot and a metatarsal pad to redistribute weight to relieve ball-of-foot discomfort. With 43% more memory foam in the forefoot for those experiencing foot discomfort or fatigue.
  Arms: Prefabricated Orthotics with metatarsal pad
Device: Aetrex L2300 Premium Memory Foam Orthotics — An Orthotic insole to be inserted into shoes. Features Aetrex Arch Support to help biomechanically align the body & help prevent common foot pain such as Plantar Fasciitis, Arch Pain and Metatarsalgia. With 43% more memory foam in the forefoot for those experiencing foot discomfort or fatigue.
  Arms: Prefabricated Orthotics without metatarsal pad.

SUMMARY:
To investigate and compare the use of a prefabricated Orthotic, with and without a metatarsal pad in decreasing pain and fear of falling in older adults.

DETAILED DESCRIPTION:
It is estimated that around 24% of community-dwelling adults over the age of 45 experience frequent foot pain. Falls and fear of falling are also significant issues in this population as both can result in avoidance of activities and decreased physical performance. In cases where fear of falling decreases physical performance and increases activity avoidance, it actually becomes a risk factor for falling itself.

Previous studies have shown that various types of Orthotic insoles improve balance and reduce lower-extremity pain in older adults. However, research which directly compares the effects of two different types of insoles is limited. Hence, this randomised control trial will investigate and compare the use of a prefabricated Orthotic, with and without a metatarsal pad, in decreasing pain and fear of falling in older adults.

This randomised control trial will be conducted over a 6-week period. The study population will include 206 participants who will be randomised into 2 groups (Group A and Group B). Participants in Group A will receive an Orthotic with a metatarsal pad and participants in Group B will receive a neutral Orthotic without the metatarsal pad. All participants will be required to continue with usual activities, using the Orthotic wherever possible for a period of 6 weeks. Participants will be asked to provide data in the form of completed surveys twice, once at the study onset and once at the end.

ELIGIBILITY:
Inclusion Criteria:

* A least 60 years of age
* Live in a community-based setting
* Are capable of ambulation
* Have some form of self-identified foot pain

Exclusion Criteria:

* Compromised skin integrity of the lower limbs
* Peripheral neuropathy and lack of sensation in the feet.
* Previous history of foot surgery and
* Inability to follow the instructions and procedures of the research protocol.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Changes in pain as assessed by a Visual Analogue Scale (VAS) | Baseline and 6 weeks
  Pain scores will be collected using the Visual Analogue Scale (VAS) as follows: Levels of pain on a 0 to 10 scale with 0 representing no pain, 2 - mild pain, 5 - moderate pain, 7 - severe pain, and 10 represents extremely severe pain. Utilization of this scale is in line with previous research [and will measure pain in the feet, ankles, knees, hips, and lower back.

SECONDARY OUTCOMES:
Changes in foot pain & functionality as assessed by the Foot Health Status Questionnaire (FHSQ) | Baseline and 6 weeks
  Foot Pain & Functionality scores will be collected using the FHSQ or Foot Health Status Questionnaire. The Foot Health Status Questionnaire is designed to assess foot pain, foot health and its relation to quality of life. The questionnaire has four domains consisting of 13 key items. The four domains are; foot pain, foot function, footwear and general foot health. The current study will only use the 2 subsections of Foot Pain and Foot Function. In these subsections, participants will be required to rate foot pain in the last week from 1 (none) to 5 (severe), how often the participant experienced different types of foot pain during the last week from 1 (never) to 5 (always), how much the participants feet interfered with everyday activities in the last week from 1 (not at all) to 5 (extremely) and overall foot health from 1 (excellent) to 5 (poor). Previous research has found the FHSQ to exhibit a strong degree of context, criterion and construct validity with high retest reliability.
Fear of falling as assessed by the Falls Efficacy Scale International (FES-I) short. | Baseline and 6 weeks
  Fear of falling will be measured using the Falls Efficacy Scale International (FES-I) short, The Falls Efficacy Scale-International (FES-I) (short) is a 7-item version of the FES-I. The questionnaire will ask participants to rate the concern about the possibility of falling when completing everyday tasks on a scale of 1 to 4 (where 1 = not at all concerned and 4 = very concerned). This version has been validated for community-dwelling older population. Furthermore, the short FES-I can predict future falls, muscle weakness, frailty and overall disability.

OTHER OUTCOMES:
Analysis of foot structure using the Gaitway scanner. | Baseline
  All the participants would undergo analysis with the Gaitway scanner. The results of the scanner will only be documented for purposes of the study and the results of the scanning will not be used to determine the Orthotic the individual participant receives.
Report how many hours, on average, the orthotics are worn each day. | 6 weeks
  Participants will be required to report how many hours, on average, the Orthotics were worn each day <4 hours, 4 to 8 hours, > 8 hours.

CONTACTS AND LOCATIONS:
Overall Officials: George Ampat, MBBS, MS, FRCS, Principal Investigator — Talita Cumi Ltd.
Locations (1):
- Talita Cumi LTD., Southport, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study, data will be fully anonymised. Only non-identifiable, anonymised data will be archived along with the publication for use of other researchers. For instance, the age, sex, and study results of participants will be archived indefinitely as a supplementary document to the publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available at the completion of the study on 31/12/2022. It will be available for other researchers indefinitely.
Access Criteria: The non-identifiable data will be openly available as a supplementary document to the publication.

REFERENCES:
- [Background] Menz HB. Chronic foot pain in older people. Maturitas. 2016 Sep;91:110-4. doi: 10.1016/j.maturitas.2016.06.011. Epub 2016 Jun 22. PMID 27451329
- [Background] Verma SK, Willetts JL, Corns HL, Marucci-Wellman HR, Lombardi DA, Courtney TK. Falls and Fall-Related Injuries among Community-Dwelling Adults in the United States. PLoS One. 2016 Mar 15;11(3):e0150939. doi: 10.1371/journal.pone.0150939. eCollection 2016. PMID 26977599
- [Background] Schoene D, Heller C, Aung YN, Sieber CC, Kemmler W, Freiberger E. A systematic review on the influence of fear of falling on quality of life in older people: is there a role for falls? Clin Interv Aging. 2019 Apr 24;14:701-719. doi: 10.2147/CIA.S197857. eCollection 2019. PMID 31190764
- [Background] Bennett PJ, Patterson C. The foot health status questionnaire (FHSQ): a new instrument for measuring outcomes of foot care. Australasian J Podiatr Med. 1998;32:55-9
- [Background] Kempen GI, Yardley L, van Haastregt JC, Zijlstra GA, Beyer N, Hauer K, Todd C. The Short FES-I: a shortened version of the falls efficacy scale-international to assess fear of falling. Age Ageing. 2008 Jan;37(1):45-50. doi: 10.1093/ageing/afm157. Epub 2007 Nov 20. PMID 18032400
- [Result] Thomas MJ, Roddy E, Zhang W, Menz HB, Hannan MT, Peat GM. The population prevalence of foot and ankle pain in middle and old age: a systematic review. Pain. 2011 Dec;152(12):2870-2880. doi: 10.1016/j.pain.2011.09.019. Epub 2011 Oct 21. PMID 22019150
- [Result] Roddy E, Muller S, Thomas E. Onset and persistence of disabling foot pain in community-dwelling older adults over a 3-year period: a prospective cohort study. J Gerontol A Biol Sci Med Sci. 2011 Apr;66(4):474-80. doi: 10.1093/gerona/glq203. Epub 2010 Nov 24. PMID 21106703
- [Result] White EG, Mulley GP. Footcare for very elderly people: a community survey. Age Ageing. 1989 Jul;18(4):276-8. doi: 10.1093/ageing/18.4.275. PMID 2816562
- [Result] Friedman SM, Munoz B, West SK, Rubin GS, Fried LP. Falls and fear of falling: which comes first? A longitudinal prediction model suggests strategies for primary and secondary prevention. J Am Geriatr Soc. 2002 Aug;50(8):1329-35. doi: 10.1046/j.1532-5415.2002.50352.x. PMID 12164987
- [Result] Mulford D, Taggart HM, Nivens A, Payrie C. Arch support use for improving balance and reducing pain in older adults. Appl Nurs Res. 2008 Aug;21(3):153-8. doi: 10.1016/j.apnr.2006.08.006. PMID 18684409
- [Result] de Morais Barbosa C, Barros Bertolo M, Marques Neto JF, Bellini Coimbra I, Davitt M, de Paiva Magalhaes E. The effect of foot orthoses on balance, foot pain and disability in elderly women with osteoporosis: a randomized clinical trial. Rheumatology (Oxford). 2013 Mar;52(3):515-22. doi: 10.1093/rheumatology/kes300. Epub 2012 Nov 28. PMID 23192905
- [Result] Perry SD, Radtke A, McIlroy WE, Fernie GR, Maki BE. Efficacy and effectiveness of a balance-enhancing insole. J Gerontol A Biol Sci Med Sci. 2008 Jun;63(6):595-602. doi: 10.1093/gerona/63.6.595. PMID 18559634
- [Result] Riskowski JL, Hagedorn TJ, Hannan MT. Measures of foot function, foot health, and foot pain: American Academy of Orthopedic Surgeons Lower Limb Outcomes Assessment: Foot and Ankle Module (AAOS-FAM), Bristol Foot Score (BFS), Revised Foot Function Index (FFI-R), Foot Health Status Questionnaire (FHSQ), Manchester Foot Pain and Disability Index (MFPDI), Podiatric Health Questionnaire (PHQ), and Rowan Foot Pain Assessment (ROFPAQ). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S229-39. doi: 10.1002/acr.20554. No abstract available. PMID 22588747
- [Result] Delbaere K, Close JC, Mikolaizak AS, Sachdev PS, Brodaty H, Lord SR. The Falls Efficacy Scale International (FES-I). A comprehensive longitudinal validation study. Age Ageing. 2010 Mar;39(2):210-6. doi: 10.1093/ageing/afp225. Epub 2010 Jan 8. PMID 20061508